CLINICAL TRIAL: NCT01159730
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Assess the Effect of Multiple Doses of VB-201 on Biomarkers
Brief Title: Study to Assess the Safety and Efficacy of Multiple Doses of VB-201 on Biomarkers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vascular Biogenics Ltd. operating as VBL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: VB-201-030
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Biomarker
MeSH Terms: interventions — 1-palmityl-2-(4-carboxybutyl)-sn-glycero-3-phosphocholine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multiple doses of VB-201 (Experimental)
  Interventions: Drug: VB-201 or Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: VB-201 or Placebo

INTERVENTIONS:
Drug: VB-201 or Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of multiple doses of VB-201 administered for 4 weeks and its efficacy on biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥18 to ≤75 years of age;

Exclusion Criteria:

* Presence of, or history of cancer, with the exception of completely excised, non-metastatic squamous cell or basal cell carcinomas of the skin;
* Has a clinically significant systemic infection (e.g., chronic or acute infection, UTI, URI) within 30 days of Day 0, or a history or presence of recurrent or chronic infection (e.g. viral infections, [including hepatitis B or C, HIV], bacterial infections, systemic fungal infections, or syphilis);
* Subjects with a history of coronary events within the last 6 months;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VBL Investigative Site, Glasgow, Scotland, United Kingdom